## INFORMED CONSENT FORM

## **Project Information**

| <b>Project Title:</b> Probing the Synergistic Effect of Pre-biotics & Iron Fortificants in Anemic Subjects | |
|---|---|
| Principal Investigator: Dr. Waqas Ahmed | |
| NCT No.: NCT03894449 | |
| <b>Date:</b> January 26, 2019 | |
| IRC Ref No.: | Organization: UVAS, Lahore |
| Address: UVAS, Outfall Road, Lahore | <b>Phone:</b> 0333-5950108 |
| Other Investigators: Abdul Momin | Organization: UVAS, Lahore |
| Address: UVAS, Outfall Road, Lahore | Phone: 0300-5332253 |

## Assalam O Alaikum!

My name is Abdul Momin Rizwan Ahmad and I am doing PhD in Food & Nutrition at the University of Veterinary & Animal Sciences, Lahore. The topic of my PhD research is "Probing the Synergistic Effect of Pre-biotics & Iron Fortificants in Anemic Subjects".

Iron deficiency anemia is one of the biggest public health problems worldwide and needs to be addressed on urgent basis. Several thousand females die of anemia each year. It has been speculated that pre-biotics when used in combination with iron fortificants may enhance the therapeutic effect against anemia but there has not been enough evidence yet.

Being an anemic adult female, you are being requested to take part in the current research study. During the 12 weeks of the research study, you will be asked to have an intake of prebiotics and iron fortificants on daily basis. You will also be required to give blood samples of 2-3 cc at the start of the study, followed by every four weeks till the completion of study, that is, 12 weeks. There are no reported side effects of pre-biotics overdose in humans as they are gut friendly substances.

The benefit which you will derive from this research study is that your anemia would be rectified by the end of the study. Moreover, there is no financial compensation for your participation in this research.

All the information gathered through this research will be kept strictly confidential and would not be revealed to anyone. Your names and identities will also be kept confidential and codes will be used to analyze the data. The results of this study may be published for scientific purposes but will not give your name or include any identifiable references to you.

You are free to choose whether or not to take part in this study. There will be no penalty or loss of benefits to which you are otherwise entitled if you choose not to participate. You will be provided with any significant new findings developed during the course of this study that may relate to or influence your willingness to continue participation.

Should you have any further questions regarding this study, you will be answered by Abdul Momin (0300-5332253).

## **AUTHORIZATION:**

I have read and understand this consent form, and I volunteer to participate in this research study. I understand that I will receive a copy of this form. I voluntarily choose to participate, but I understand that my consent does not take away any legal rights in the case of negligence or other legal fault of anyone who is involved in this study.

| Name of participant: |
|--------------------------------------------|
| Signature/Thumb Impression of participant: |
| Date: |
| Name of person obtaining consent: |
| Signature of person obtaining consent: |
| Date: |
| Signature of Principal Investigator: |
| Date: |